CLINICAL TRIAL: NCT04230512
Title: Hybrid Electrical-Mechanical Pump for Vacuum Suspension of Prosthetic Sockets
Brief Title: Hybrid Pump Technology
Acronym: HIPPI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A3090-R; RX003090-01A2 (Other Grant/Funding Number: Dept Veterans Affairs)
Record Dates: First submitted 2019-11-15; First posted 2020-01-18 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Amputation
Keywords: Amputation; Prosthesis; Gait; Leg

STUDY DESIGN:
Intervention Model Description: Randomly assigned conditions of pump function to characterize the effects of added movement on socket-reaction torques
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Locked (Experimental): The prototype mechanical system is locked from compressing
  Interventions: Other: Pump prototype
- Unlocked (Experimental): The prototype mechanical system is free to compress normally
  Interventions: Other: Pump prototype

INTERVENTIONS:
Other: Pump prototype — Effects of pump function on gait

SUMMARY:
Prostheses can be suspended from the amputated limb using a variety of techniques, such as straps and suction. Suspending the prosthesis by creating a vacuum between the prosthetic socket and limb using a pump has benefits over other techniques including improved limb health and mobility. A new pump design will be tested by prosthesis users in the laboratory to verify its functionality during walking.

DETAILED DESCRIPTION:
Human subject testing will involve a cross-sectional, repeated measures study consisting of a single 3 hour visit wherein participants will initially stand and then continuously walk at their self-selected speed for ten minutes on a level treadmill with the prototype under two randomly presented conditions of the mechanical system: 1) fully functional, and 2) locked to restrict axial displacement. After written informed consent is obtained, information on socket comfort and mobility capability will be collected. A load-cell will be installed proximal to the prototype and in-line with the prosthesis to measure instantaneous socket-reaction moments.

ELIGIBILITY:
Inclusion Criteria:

* Ability to stand quietly and walk for 10 minutes continuously without an assistive device (e.g. cane or walker) and without undue fatigue or health risks
* Pre-classified clinically to be at least a limited community ambulator of Medicare Functional Classification Level (K)2
* Residual limb in good health
* At least six months experience with a definitive prosthesis that utilizes vacuum assisted suspension

Exclusion Criteria:

* Pathologies aside from amputation or taking medicine that would influence walking or balance
* Poor prosthetic fit or poor residual limb sensation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-04-04 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Socket-reaction moments | Immediate
  Moments (torques) generated at the prosthetic socket end during walking

SECONDARY OUTCOMES:
Socket Comfort | Immediate
  Comfort of the prosthetic socket
Perceived mobility capability | Immediate
  Mobility capability as reported by the participant

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Major, PhD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No